CLINICAL TRIAL: NCT05524974
Title: Clinical Efficacy of Carrelizumab, Apatinib Mesylate, Albumin Paclitaxel Combined With Oxaliplatin and S-1 in Neoadjuvant Treatment of Locally Advanced Gastric Cancer With Different Genotypes--A Prospective, Multi-center, Randomized Controlled Study
Brief Title: Clinical Study of Camrelizumab, Apatinib Mesylate and Nab-paclitaxel Combined With Oxplatin and S-1 in the Neoadjuvant Treatment of Locally Advanced Gastric Cancer With Different Genotypes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director of gastric surgery, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Arise-FJ-G006
Record Dates: First submitted 2022-08-10; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Locally Advanced Gastric Cancer
MeSH Terms: interventions — camrelizumab; Oxaliplatin; S 1 (combination); apatinib; Taxes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Camrelizumab combined with Oxplatin and S-1 for Immune Genotypes (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Oxaliplatin; Drug: S1
- Oxplatin and S-1 for Immune Genotypes (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: S1
- Apatinib Mesylate combined with Oxplatin and S-1 for Mesenchymal Genotypes (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: S1; Drug: Apatinib Mesylate
- Oxplatin and S-1 for Mesenchymal Genotypes (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: S1
- Nab-paclitaxel combined with Oxplatin and S-1 for Classic Genotypes (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: S1; Drug: Nab paclitaxel
- Oxplatin and S-1 for Classic Genotypes (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: S1
- Oxplatin and S-1 for Metabolic Genotypes (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: S1

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab One course will last 21 days. Given once every 3 weeks at a dose of 200 mg.
  Arms: Camrelizumab combined with Oxplatin and S-1 for Immune Genotypes
Drug: Oxaliplatin — Oxaliplatin for Injection 135mg/m2 /per day，ivgtt，in day1. Given once every 3 weeks.
Drug: S1 — S-1 was calculated according to body surface area , P.O., bid, d1-d14. And the dosage according body surface area:<1.25m2, 40mg every time;1.25-1.5m2,50mg every time; >1.5m2, 60mg every time
Drug: Apatinib Mesylate — Apatinib One course will last 21 days.Oral administration at a dose of 250 mg everyday.
  Arms: Apatinib Mesylate combined with Oxplatin and S-1 for Mesenchymal Genotypes
Drug: Nab paclitaxel — nab-paclitaxel One course will last 21 days. Given twice every 3 weeks at a dose of 260 mg/m2 in day 1 and day 8.
  Arms: Nab-paclitaxel combined with Oxplatin and S-1 for Classic Genotypes

SUMMARY:
To evaluate the clinical efficacy of camrelizumab, apatinib Mesylate and nab-paclitaxel combined with oxplatin and S-1 in the neoadjuvant treatment of locally advanced gastric cancer with different genotypes

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years, all sex；
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by histology or cytology；
3. CT/MRI,PET-CT or laparoscopic exploration were used to confirm the diagnosis of gastric cancer staging as cT2-4a and/or N+ and M0 before operation.；
4. measurable lesions at least should be detected by CT/MRI examination in accordance with the RECIST1.1.（CT scan of tumor lesion length≥10mm，CT scan short diameter of lymph node≥15mm，scan slice thickness 5mm）;
5. ECOG（Eastern Cooperative Oncology Group）PS（Performance Status）:0-1 scores;
6. the expected survival time is more than 12 weeks;
7. the main organ function is normal, which should meet the following criteria: （1）(1)blood routine examination standards should be met（no blood transfusion within 14 days）

   1. HB≥100g/L，
   2. WBC≥3×109/L
   3. ANC≥1.5×109/L，
   4. PLT≥100×109/L； （2）biochemical examination shall comply with the following criteria：

   <!-- -->

   1. BIL <1.5normal upper limit（ULN），
   2. ALT和AST<2.5ULN，GPT≤1.5×ULN；
   3. serum Cr≤1ULN，creatinine clearance rate>60ml/min（Cockcroft-Gault formula）
8. women of childbearing age must have a pregnancy test in 7 days before entering the group (in serum), and the results were negative, and willing to use appropriate contraception during the study period and the last 8 weeks after giving drug; men should have the surgical sterilization, or adopt the appropriate contraceptive methods during the test and the last 8 weeks after giving drug.；
9. No other clinical studies were conducted before and during the treatment； participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up.

Exclusion Criteria:

1. Previous history of chemotherapy, radiotherapy, targeted drug therapy or immunotherapy
2. Patients with contraindications for surgical treatment and chemotherapy or whose physical condition and organ function do not allow for major abdominal surgery；
3. patients with metastasis；
4. Having any active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Patients with vitiligo or cured childhood asthma/allergies who did not need any intervention in adulthood were excluded; Autoimmune hypothyroidism treated with a stable dose of thyroid replacement hormone; Type 1 diabetes with stable doses of insulin；
5. A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation；
6. Accompanied by serious heart, lung, liver, kidney disease; Have nerve, mental disease; Jaundice or obstruction of the digestive tract with severe infection；
7. pregnant or lactating women；
8. The blood pressure of patients with hypertension cannot be reduced to the normal range by the antihypertensive drugs (systolic pressure >140 mmHg, diastolic pressure >90 mmHg)；
9. With Ⅰ magnitude of coronary heart disease, arrhythmia (including QTc protracted between male > 450 ms, women > 470 ms) and cardiac insufficiency；
10. Patients have a clear tendency with gastrointestinal bleeding, including the following situation: local active ulcerative lesions, and fecal occult blood (+ +); with melena and hematemesis history in 2 months; and patients with fecal occult blood (+) and coagulation dysfunction (INR(international normalized ratio)>1.5, APTT(activated partial thromboplastin time)>1.5 ULN), with bleeding tendency;；
11. Subjects have failed to control good cardiovascular clinical symptoms or disease, including but not limited to: such as: (1) the NYHA class II heart failure or above (2) unstable angina pectoris (3) MI occurred within 1 year (4) have clinical significance of supraventricular or ventricular arrhythmias without clinical intervention on or after clinical intervention is still poorly controlled；
12. History of interstitial lung disease (except radiation pneumonia without hormone therapy), and history of non-infectious pneumonia；
13. Patients are positive of urine protein (urine protein detection 2+ or above, or 24 hours urine protein quantitative >1.0g)；
14. A person who has previously been allergic to any component of the drug in this study； The researchers consider those who were not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 4 months
  Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST

SECONDARY OUTCOMES:
R0 resection rate | 4 months
  The surgical procedure was total or subtotal gastrectomy with 3 weeks after total neoadjuvant therapy.
Disease control rate | 4 months
1-year and 3-year OS/DFS | 1 and 3 years
adverse event | 3 years
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
overall postoperative morbidity rates | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery.
30 days mortality rates | 30 days
  Defined as the event observed within 30 days after surgery.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
The prediction performance of Exosome contents (including proteins, nucleic acids) | 3 years
  Exosomes were isolated using a Backman Optima XPN-100 instrument. The exosomes morphology was characterized using a HT7700 transmission electron microscope (Hitachi, Co. Ltd., Japan). Fluorescent spectra were recorded using a F96 Pro fluorospectrophotometer (Shanghai Lengguang Technology). The concentration and size distribution of the exosomes were quantified using nanoparticle tracking analysis (NanoSight NS 300, Malvern Instrument). The obtained results were subjected to biostatistical analysis, such as heat map generation, ROC curve establishment, and confusion matrix.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, phD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China